CLINICAL TRIAL: NCT01163656
Title: A Prospective Comparison of the Glidescope Cobalt to Standard Direct Laryngoscopy in Infants
Brief Title: Comparing Use of the Glidescope Cobalt to Direct Laryngoscopy in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-007533
Record Dates: First submitted 2010-07-13; First posted 2010-07-16 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Intubation
Keywords: Neonate; Laryngoscopes
MeSH Terms: interventions — Intubation, Intratracheal; Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Laryngoscopy (Active Comparator): Laryngoscopy will be performed with the randomized device, which will be the Miller Laryngoscope.
  Interventions: Device: Miller Laryngoscope
- Glidescope Cobalt Video Laryngoscopy (Active Comparator): Laryngoscopy will be performed with the randomized device, which will be the Glidescope Cobalt Video Laryngoscope.
  Interventions: Device: Glidescope Cobalt Video Laryngoscopes

INTERVENTIONS:
Device: Miller Laryngoscope — Device is used to facilitate tracheal intubation.
  Other Names: tracheal intubation; laryngoscopy; direct laryngoscopy
  Arms: Direct Laryngoscopy
Device: Glidescope Cobalt Video Laryngoscopes — The laryngoscope design with the integration of video technology into the laryngoscope blade.
  Other Names: Glidescope Cobalt Video Laryngoscopy; Video Laryngoscopy
  Arms: Glidescope Cobalt Video Laryngoscopy

SUMMARY:
The investigators seek to prospectively compare intubation with the Glidescope Cobalt to Direct Laryngoscopy (DL) in infants.

DETAILED DESCRIPTION:
We seek to study the intubation characteristics of a new video laryngoscope, the Glidescope Cobalt in children less than or equal to 1 yr of age. This evaluation would provide insight as to the efficacy of this device in facilitating intubation in infants.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo elective surgery at CHOP
2. American Society of Anesthesiologists (ASA) Physical Status I or II
3. Anesthetic plan requiring tracheal intubation with a neuromuscular relaxant
4. Parental/guardian permission (informed consent). Subjects will be too young to understand the study procedures and therefore assent will not be sought. -

Exclusion Criteria:

1. At known or anticipated high risk for aspiration pneumonia
2. Known or predicted difficult intubation as assessed by the clinical attending anesthesiologist
3. Emergency surgical procedure
4. Patients with preoperative airway pathology or stridor -

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fiadjoe, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy infants under the age of 12 months undergoing elective surgery requiring tracheal intubation were eligible.
Pre-assignment Details: Any subject was excluded from participation if they were known or suspected to be a difficult intubation or if they required a rapid-sequence intubation.
Groups:
- Direct Laryngoscopy Approach; Glidescope Videoscope Approach: Subjects were randomly assigned to an arm.
Period: Overall Study
Arm/Group | Direct Laryngoscopy Approach | Glidescope Videoscope Approach
Started | 33 | 33
Completed | 30 | 30
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Laryngoscopy Approach | Glidescope Videoscope Approach | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 33 | 66
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.425 (0.275) | 0.492 (0.283) | 0.459 (0.279)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 20 | 28 | 48
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Time to Tracheal Intubation
Description: The amount of time it takes the anesthesiologist to insert a breathing tube using one of two methods, either by direct laryngoscopy or using the Glidescope Cobalt Video system.
Time Frame: Measured the time of the randomized device past the teeth/gums until its removal after intubation as the time to intubation.
Measure: Median (95% Confidence Interval); unit: seconds
Arm/Group | Direct Laryngoscopy Approach | Glidescope Videoscope Approach
Number analyzed (Participants) | 30 | 30
seconds | 21.4 [9.5 to 66.1] | 22.6 [13.3 to 61.0]

ADVERSE EVENTS:
Arm/Group | Direct Laryngoscopy Approach | Glidescope Videoscope Approach
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No